CLINICAL TRIAL: NCT00168545
Title: Non-specific Effects of Vaccines - In Search of the Immunological Background
Brief Title: Immunology of Non-specific Effects of Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: Novo Nordisk A/S (Industry); Fonden til Lægevidenskabens Fremme (Other); Danish Council for Development Research (Other); Medical Research Council Unit, The Gambia (Other); Leiden University Medical Centre, DEPT of Parasitology, Leiden Holland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NOVO-2624-Twodose2_immunology; NOVO-2624; LÆGEVIDENSKABENS FREMME-2623
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2006-09

CONDITIONS: Measles; Diphtheria; Tetanus; Pertussis
Keywords: Non-specific effects of vaccines; Immunology; Cytokines; Infant mortality; Child mortality; Mortality; Morbidity; Diphtheria-tetanus-pertussis vaccine; Measles vaccine; Measles; Immunisation; Low income country; Guinea-Bissau; Bandim Health Project; Immunology of measles and DTP vaccination
MeSH Terms: conditions — Measles; Diphtheria; Tetanus; Whooping Cough; Infant Death | interventions — Measles Vaccine

INTERVENTIONS:
Biological: Measles vaccine

SUMMARY:
OBJECTIVES

* General: To investigate the immunological background for the non-specific effects of diphtheria-tetanus-pertussis (DTP) and measles vaccines on child mortality
* Specific: Examine the cytokine responses and possible association with morbidity in a study of DTP vaccinated children who will be randomised to receive a measles vaccine or no vaccine at 4½ months of age. (All children will receive a measles vaccine at 9 months of age)

DETAILED DESCRIPTION:
Non-specific effects of vaccines The idea of vaccines having non-specific effects was first proposed in 1991 from a study in Senegal, West Africa. It was discovered that children receiving high-titre measles vaccine (HT) at 6 months of age had higher mortality than children who received the standard titre measles vaccine (STD) at 9 months of age. The difference was found only for girls. A study from Haiti confirmed the effect. Since children vaccinated with HT had lower mortality than their equivalents who had not received any measles vaccine, the difference in mortality between recipients of HT vaccine and STD vaccine was explained by a non-specific beneficial effect of the STD measles vaccine rather than a harmful effect of the HT vaccine. The non-specific beneficial effect of STD measles vaccine on child mortality has been reconfirmed in many data-sets.

Also the BCG vaccine is associated with striking effects on child mortality reducing mortality by about 50%. Further, among BCG vaccinated children, having a BCG scar or a positive tuberculin reaction was associated with about 55% lower mortality in the following 12 months than among children who had a negative tuberculin reaction or who did not have a BCG scar.

The effect of OPV is difficult to separate from the effects of BCG and DTP vaccines since OPV is normally given together with these vaccines. There have, though, been some periods without DTP in Bissau due to global shortage of vaccines, and we have compared the case fatality at the hospital for children who received only OPV and children who received both the prescribed OPV and DTP. Children having received OPV had 3-fold lower mortality than children having received both vaccines. Data from an OPV vaccination campaign that took place in Guinea-Bissau also suggested a non-specific beneficial effect for the recipients. Further, studies from Chile and the Soviet Union have suggested that OPV had a beneficial effect on mortality and morbidity.

In contrast, DTP, HBV and inactivated polio vaccine (IPV) seem to exert a non-specific detrimental effect on child mortality, although the findings on DTP were considered controversial by a recent review. Current studies indicate that the negative effect of DTP may be neutralized by a subsequent measles vaccination. It is striking that all the vaccines with a non-specific beneficial effect are live, whereas the vaccines with an apparently harmful effect are killed. Results from animal studies have shown that attenuated live vaccines tend to induce a Th1 response and offer better protection against severe disease than the corresponding inactivated vaccines, which tend to induce a Th2 response. So far, very few studies have examined whether these effects differ between male and female animals. One study reported that BCG-vaccinated female mice were better protected against malaria parasites than male mice (31). There is therefore an urgent need to conduct studies that can help uncover the immunology behind the non-specific effects.

Sex-specific effects All epidemiological studies carried out so far confirms the observation that non-specific effects are sex-specific. Live vaccines (measles, BCG, OPV) have a beneficial effect that is particularly good for girls whereas inactivated vaccines (DTP, HBV, IPV) have a negative effect for girls. To date, there are no immunological studies which have examined whether routine vaccines affect the immune system differently for boys and girls.

We thus propose to study, in a randomised controlled trial of measles vaccination taking place in Guinea-Bissau, the immunology of non-specific effects of vaccination, and their interaction with sex. Specifically, among children who have received the 3 recommended doses of DTP, we will be able to compare the cytokine and antibody profiles of children who receive an early dose of measles vaccine at 4½ months of age with children who receive no additional vaccine at this age.

ELIGIBILITY:
Inclusion Criteria: A sub-cohort of children participating in the study "MEASLES VACCINATION IN GUINEA-BISSAU. STRATEGIES TO REDUCE DISEASE BURDEN AND IMPROVE CHILD SURVIVAL", protocol ID: RUF-91134-2601-Twodose2.

Exclusion Criteria: Severe illness

Ages: 4 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400
Dates: Start 2006-01; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Cytokine levels in the randomised groups

CONTACTS AND LOCATIONS:
Overall Officials: PETER AABY, MSc, Dr Med, Study Director — Bandim Health Project; MAY-LILL GARLY, PHD, DTM&H, Principal Investigator — Bandim Health Project
Locations (1):
- Bandim Health Project, Bissau, Apartado 861, Guinea-Bissau

REFERENCES:
- [Derived] Jensen KJ, Sondergaard M, Andersen A, Sartono E, Martins C, Garly ML, Eugen-Olsen J, Ullum H, Yazdanbakhsh M, Aaby P, Benn CS, Erikstrup C. A randomized trial of an early measles vaccine at 4(1/2) months of age in Guinea-Bissau: sex-differential immunological effects. PLoS One. 2014 May 16;9(5):e97536. doi: 10.1371/journal.pone.0097536. eCollection 2014. PMID 24835247
- See also: Statens Serum Institut, Denmark — http://www.ssi.dk